CLINICAL TRIAL: NCT05999838
Title: High-resolution Chest CT Visual Scoring, Spirometry and Health Related Quality of Life in Evaluating Severity of Interstitial Lung Disease Patients
Brief Title: HR Chest CT Visual Scoring, Spirometry and Health Related Quality of Life in Evaluating Severity of ILD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Wageeh Fahim, Doctor, Assiut University
Other Study IDs: HR chest CT spirometry ILD
Record Dates: First submitted 2023-07-11; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HRCT chest visual scoring — CT-based semi-quantitative scoring will be calculated according to number of lung segments affected on both sides.
  The finding on each segment will be given a score from 1 to 4 as follows:
  1. for ground glass opacities.
  2. for reticulations and fibrotic changes.
  3. for bronchiectatic changes.
  4. for honeycombing and sub-pleural cysts.
  Other Names: spirometry

SUMMARY:
To establish a simplified approach for assessment of severity of interstitial lung disease by evaluating the relationship between HRCT findings, the clinical severity score,spirometry and quality of life.

DETAILED DESCRIPTION:
The interstitial lung diseases are a group of parenchymal pulmonary disorders that affect the interstitium causing progressive fibrosis of lung tissue. These disorders characterized by dyspnea aggravated by exertion . This group of diseases is associated with substantial morbidity and mortality. Thus, a multi-disciplinary approach including clinical, pathological, and radiological correlation is required to reach accurate assessment. The high-resolution computed tomography [HRCT] images of the chest are considered the main platform for the diagnostic approach .High-resolution CT (HRCT) scans offer the possibility of measuring disease severity more accurately and sensitively by focusing on fibrotic changes. HRCT images illustrate the presence and extent of parenchymal abnormalities including: reticular opacities, ground-glass opacities, traction bronchiectasis and honeycombing. Most patients with suspected ILDs are likely to undergo complete Pulmonary Function Testing. Usually there is restrictive pulmonary function with decreased TLC (Total Lung Capacity) , FVC (Forced Vital Capacity), FEV1 (Forced Expiratory Volume in One Second) and a normal or increased FEV1/FVC ratio.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted at Chest Department or presented to our out patient clinic with clinical diagnosis of Interstitial Lung Diseases among both sexes

Exclusion Criteria:

* patients under 18 years old.
* pregnant patients.
* patients with a history of previous lung resections.
* presence of bronchial carcinoma or lobar consolidation.
* patients contraindicated to perform pulmonary function will be excluded.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted at Chest Department or presented to our out patient clinic with clinical diagnosis of Interstitial Lung Diseases
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Correlation of visual based scoring system of HRCT and pulmonary function test. | 1 year

SECONDARY OUTCOMES:
assessment of ILDs patients quality of life and correlation with HRCT finding and PFTs. | 1 year